CLINICAL TRIAL: NCT06901817
Title: A Multicenter, Prospective, Phase II Study on Intraventricular Injection of Pemetrexed Combined with Nivolumab Via an Ommaya Reservoir for the Treatment of Refractory Non-squamous Non-small Cell Lung Cancer (NSCLC) with Leptomeningeal Metastases in Previously Treated Patients
Brief Title: A Study of the Safety and Efficacy of Pemetrexed Combined with Nivolumab Via Intraventricular Injection for the Treatment of Refractory Non-squamous Non-small Cell Lung Cancer with Leptomeningeal Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Principal Investigator, Fan Min, Vice president of Department of Radiation Oncology, Shanghai Cancer Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC20240710
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraventricular Pemetrexed combined with Nivolumab (Experimental): Patients with leptomeningeal metastases from refractory non-squamous non-small cell lung cancer will receive Pemetrexed and Nivolumab vis Ommaya reservoir.
  Interventions: Drug: Intraventricular Pemetrexed; Drug: Intraventricular Nivolumab; Drug: Intraventricular Dexamethasone

INTERVENTIONS:
Drug: Intraventricular Pemetrexed — Intraventricular injection of 30 mg pemetrexed via Ommaya reservoir, once every 4 weeks until disease progression.
Drug: Intraventricular Nivolumab — Intraventricular injection of 40 mg nivolumab via Ommaya reservoir, once every 4 weeks until disease progression.
Drug: Intraventricular Dexamethasone — Intraventricular injection of 5mg/2ml pemetrexed via Ommaya reservoir before injection of pemetrexed and nivolumab.

SUMMARY:
The goal of this clinical trial is to learn if the intraventricular injection of Pemetrexed and Nivolumab works to treat refractory non-squamous non-small cell lung cancer with leptomeningeal metastases. The main questions to answer are:

* Is the combination of Pemetrexed and Nivolumab safe to inject?
* How effective is the combination in disease control?

Participants will：

* Intrathecal injection of 30 mg pemetrexed via Ommaya reservoir, once every 4 weeks until disease progression;
* Intrathecal injection of 40 mg nivolumab via Ommaya reservoir, once every 4 weeks until disease progression;
* Before each intrathecal administration, a preliminary intrathecal injection of dexamethasone, 5 mg/2 mL, is given.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent form and are willing to complete the study according to the protocol;
* Patients must have radiographic and/or cerebrospinal fluid cytology evidence of leptomeningeal disease (LMD). The diagnosis of non-small cell lung cancer must be confirmed, based on histological and/or cytological diagnosis.
* Patients must have an ECOG performance status score of ≤ 2.
* Patients may use steroids to control symptoms related to the central nervous system, but the dose must be ≤ 4 mg of dexamethasone (or equivalent dose) within 24 hours. The patient's neurological symptoms should remain stable for at least 7 days, or they are reducing the dose of steroids. Physiological replacement doses for adrenal insufficiency are allowed.
* Patients who have received brain and/or spinal radiotherapy, including whole-brain radiation, stereotactic radiosurgery, or SBRT, can be enrolled, but must have completed radiation therapy at least 7 days before starting treatment.
* Patients who have received approved systemic treatments may continue the systemic treatment chosen by the researcher. Concurrent use of other drugs for intrathecal treatment is not allowed. For patients who have received other systemic treatments, the minimum washout periods are as follows:

  1. Patients who have received intrathecal treatment must have had their last treatment at least 7 days before starting the study treatment.
  2. Patients who have received systemic chemotherapy must have had their last treatment at least 14 days before starting the study treatment.
  3. Patients who have received approved systemic immunotherapy (such as anti-PD-1, anti-CTLA4) must have had their last treatment at least 2 weeks before starting the study treatment.
  4. Patients who have received any other investigational drugs must have had their last treatment at least 14 days before starting the study treatment.
* Age ≥ 18 years.
* Able to provide written informed consent, including compliance with the requirements and restrictions listed in the consent form.
* Patients must have the organ and bone marrow function defined in Table 1 below.
* No contraindications to the installation of an Ommaya reservoir.
* Criteria for refractory leptomeningeal metastasis:

  1. Failed first- or second-generation TKI treatment, T790M mutation-negative;
  2. Failed third-generation TKI treatment;
  3. EGFR gene mutation-negative, failed first-line treatment.

Exclusion Criteria:

* Patients who require a VP shunt due to increased intracranial pressure.
* Patients must not have active autoimmune diseases requiring systemic treatment in the past two years (i.e., using disease-modifying agents, corticosteroids, or immunosuppressive drugs). Alternative therapies (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered forms of systemic treatment.
* Subjects who need systemic treatment within 14 days prior to administration of the study drug, including the use of corticosteroids (>4 mg daily dexamethasone equivalent dose) or other immunosuppressive drugs. Inhaled or topical steroids and adrenal replacement therapy at a daily replacement dose >10 mg prednisone equivalent are allowed in the absence of active autoimmune diseases.
* Patients who have previously received PD-1 and/or anti-CTLA-4 therapy are eligible, unless they are experiencing > grade 2 side effects from such treatments. Ongoing physiological replacement doses for adrenal and thyroid insufficiency are allowed in the protocol.
* Patients currently receiving experimental anti-cancer drugs (co-treatment with approved targeted therapies is permitted).
* Patients with a history of other malignancies are eligible if they have appropriately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other cancers with no evidence of disease for more than 5 years.
* Participation in another clinical trial within 30 days prior to randomization, receiving investigational drugs and any concomitant treatments containing investigational drugs.
* Immunodeficiency, HIV infection;
* Severe dysfunction of the heart, lungs, liver, or kidneys;
* Uncontrolled infection or active infection;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 30 days
  Per CTCAE version 4.0

SECONDARY OUTCOMES:
objective response rate (ORR) | 1 year
  LM objective response rate (ORR) is defined as the proportion of patients with at least one objective response in LM, using a combined approach taking into account radiographic, neurologic and cytologic assessments based on RANO-LM.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No